CLINICAL TRIAL: NCT04634812
Title: A Phase 1, Open-label, Study of the Absorption, Metabolism, and Excretion of [14C]-KBP-5074 Following a Single Oral Dose in Healthy Male Subjects
Brief Title: Mass Balance Study of KBP-5074 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: KBP Biosciences (Industry)
Collaborators: Covance (Industry)
Responsible Party: Sponsor
Organization: Novo Nordisk A/S (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: KBP5074-1-007
Record Dates: First submitted 2020-11-12; First posted 2020-11-18 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Healthy
Keywords: Healthy Male Subjects; KBP-5074
MeSH Terms: interventions — KBP-5074

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [14C]-KBP-5074 (Experimental)
  Interventions: Drug: KBP-5074

INTERVENTIONS:
Drug: KBP-5074 — a single oral dose of [14C]-KBP-5074

SUMMARY:
This is a Phase 1, open-label, nonrandomized, single-dose mass balance and metabolite identification study in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Males, of any race, between 18 and 55 years of age, inclusive, at screening.
2. Body mass index between 18.0 and 32.0 kg/m2, inclusive, at screening.
3. In good health, determined by no clinically significant findings from medical history, physical examination (assessed only at check-in), 12-lead ECG, vital sign measurements, and clinical laboratory evaluations (congenital nonhemolytic hyperbilirubinemia [eg, suspicion of Gilbert's syndrome based on total and direct bilirubin] is not acceptable) at screening and check-in as assessed by the investigator (or designee).
4. History of a minimum of 1 bowel movement per day.

Exclusion Criteria:

1. Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, psychiatric, or other disorder, as determined by the investigator (or designee).
2. History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs (uncomplicated appendectomy and hernia repair will be allowed; cholecystectomy will not be allowed).
3. Positive urine drug screen, including cotinine, at screening; positive alcohol test result or positive urine drug screen, including cotinine, at check-in.
4. Use of any drugs or substances known to be strong or moderate inhibitors or inducers of cytochrome P450 (CYP)3A4 or P-glycoprotein substrates within 30 days prior to study drug administration. Medications will be reviewed by the medical monitor to determine acceptability for the study.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2020-12-03 (Actual); Primary Completion 2020-12-23 (Actual); Study Completion 2020-12-23 (Actual)

PRIMARY OUTCOMES:
Mass Balance of KBP-5074 | up to 240 hours postdose
  Percentage of total radioactivity recovered in urine and feces following a single dose [14C]-KBP-5074
Pharmacokinetic Parameter: Area under the concentration-time curve from time 0 to infinity (AUC0-∞) | up to 216 hours postdose
  Area under the concentration-time curve from time 0 to infinity (AUC0-∞) - Plasma
Pharmacokinetic Parameter: Area under the plasma concentration time curve from time zero to time of last quantifiable concentration (AUC0-tlast) | up to 216 hours postdose
  Area under the plasma concentration time curve from time zero to time of last quantifiable concentration (AUC0-tlast) - Plasma
Pharmacokinetic Parameter: Time of the maximum observed concentration (Cmax) | up to 216 hours postdose
  Time of the maximum observed concentration (Cmax) - Plasma

SECONDARY OUTCOMES:
Metabolite radioprofiling and identification in plasma, urine and feces | up to 240 hours postdose
  Select plasma, urine, and fecal samples will be processed and subject to metabolite analysis by LC/MS & LC/MS/MS using high-resolution mass spectrometry.

CONTACTS AND LOCATIONS:
Overall Officials: James McCabe, Study Director — KBP Biosciences
Locations (1):
- Covance Clinical Research Unit Inc., Madison, Wisconsin, United States